CLINICAL TRIAL: NCT03918733
Title: Comparative Evaluation of Clinical and Radiographic Outcome of Nonsurgical Retreatment and Endodontic Surgery of Root Filled Teeth"
Brief Title: Comparision of Non Surgical Retreatment and Endodontic Surgery of Failed Root Canal Treated Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: usha yadav
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Root Canal Therapy; Periapical Periodontitis
Keywords: retreatment; endodontic surgery; nonsurgical endodontic retreatment
MeSH Terms: conditions — Periapical Periodontitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical treatment (Experimental): surgical treatment of failed root canal treated teeth following secondary root canal treatment.
  Interventions: Procedure: surgical treatment
- Non surgical retreatment (Experimental): Non surgical retreatment of failed root canal treated teeth
  Interventions: Procedure: Non surgical retreatment

INTERVENTIONS:
Procedure: surgical treatment — surgical treatment will be done of failed root canal treated teeth
  Arms: surgical treatment
Procedure: Non surgical retreatment — Non surgical retreatment will be done.
  Arms: Non surgical retreatment

SUMMARY:
To the best of our knowledge, only two studies are available which have provided a direct comparison between outcome of nonsurgical retreatment and endodontic surgery. The results of the two studies are contradictory in nature. Two systematic reviews conducted to explore the issue also could not draw any definitive conclusions and suggested that further research is necessary to find out effects of surgical versus nonsurgical approach. Considering the very limited amount of data on this pertinent topic, there is apparent need of high quality randomized controlled studies to further investigate the difference in outcome between nonsurgical retreatment and endodontic surgery.

DETAILED DESCRIPTION:
TITLE: Comparative evaluation of clinical and radiographic outcome of nonsurgical retreatment and endodontic surgery of root filled teeth.

RATIONALE: To the best of our knowledge, only two studies are available which have provided a direct comparison between outcome of nonsurgical retreatment and endodontic surgery. The results of the two studies are contradictory in nature. Two systematic reviews conducted to explore the issue also could not draw any definitive conclusions and suggested that further research is necessary to find out effects of surgical versus nonsurgical approach. Considering the very limited amount of data on this pertinent topic, there is apparent need of high quality randomized controlled studies to further investigate the difference in outcome between nonsurgical retreatment and endodontic surgery.

AIM AND OBJECTIVES: Evaluate and compare the clinical and radiographic outcomes of nonsurgical endodontic retreatment and endodontic surgery.

SETTING: Study subjects should be recruited from the Post Graduate Department of Conservative Dentistry and Endodontics, PGIDS, Rohtak, Haryana.

STUDY DESIGN: Prospective randomized study

Method: Patients with above inclusion criteria will be selected and randomly allocated to one of the two study groups ( nonsurgical retreatment , endodontic microsurgery ). Root canal retreatment will be performed according to standard protocol. Surgical procedures will be carried out under operating microscope with 8 × 16 magnification by following standardized treatment methods.

Outcome measures: Follow up will be done every 3 months till 12 month period to assess clinical and radiographic success of nonsurgical retreatment and endodontic microsurgery. Clinical success will be assessed by absence of pain and tenderness to palpation/ percussion, absence of sinus or any associated soft tissue swelling, tooth mobility of grade-I or less, and no deterioration in periodontal probing depth. Radiographic success will be assessed by the criteria followed by Rud et al. (1972) and Molven et al. (1987). Intensity of pain will be assessed using Visual Analog Scale. Pain intensity will be recorded at different intervals (preoperatively, after 6 hours, 12 hours, 18 hours, 1day, 2 days, 3 days, 4 days, 5 days, 6 days and 7 days). Intake of analgesic will also be recorded.

Statistical Analysis: The data gathered will be analyzed using suitable statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* • Patient willingness to participate in the study.

  * Previously root filled Permanent teeth with post-treatment apical periodontitis requiring treatment.
  * Radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm2).
  * Failure of previous root canal treatment will be determined based on clinical and radiographic examinations.
  * Patient's age more than 18 years.

Exclusion Criteria:

* Positive history of antibiotic use within past three months of the treatment.
* Positive history of analgesic use within the past 7 days.
* Procedural errors in previous root canal treatment which are not manageable.
* Patients who are pregnant, diabetic, having human immunodeficiency virus infection or other immunocompromising conditions, had serious medical illness or requiring antibiotic premedication.
* Patients with unrestorable lesions, fractures involving the periodontium, and/or periodontal pockets ≥ 4mm deep or having marginal or furcal bone loss due to periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic success | Baseline to one year
  Follow up will be done every 3 months till 12 months. scoring of each tooth will be done according to criteria followed by Rud et al (1972) and Molven et al (1987)
  1. Complete healing, defined by re-establishment of the lamina dura
  2. Incomplete healing (scar tissue)
  3. Uncertain healing
  4. Unsatisfactory healing (failure)

CONTACTS AND LOCATIONS:
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India